CLINICAL TRIAL: NCT01476514
Title: Effects of Mutations of the Glycine Gene Associated With Hyperekplexia on Central Pain Processing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Pascal H. Vuilleumier, MD, University Hospital Bern, Switzerland
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 131/11; SPUM no. 33CM30_124117
Record Dates: First submitted 2011-11-02; First posted 2011-11-22 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Hyperekplexia
Keywords: Hyperekplexia; Pain modulation; Glycine receptors; Hyperalgesia; Spinal inhibitory interneurons
MeSH Terms: conditions — Hyperekplexia; Hyperalgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In the setting of comparing patients with a genetic mutation and healthy volunteers blinding of the PI would demand a substantial increase in co-workers (i.e. recruitment, selection of age-and sex matched volunteers), reason why no blinding was chosen.
  Affected patients will be compared to age and sex matched volunteers, recruited after completion of testing 23 hyperekplexia patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The testing will be the same for healthy volunteers and patients with a mutations in the glycine channel.

SUMMARY:
Mutations in genes affecting pain transmission start to be known, the investigators are investigating a mutation in a glycine channel, which has an influence on pain modulation. Pain modulation is the ability of the central nervous system to enhance or diminish the sensation of pain. The investigators therefore will test patients and healthy volunteers with quantitative sensory tests, basically determining the point at which a stimulation just starts to induce pain. These tests are reliable and permit a direct comparison between healthy volunteers and patients with the affected glycine gene.

DETAILED DESCRIPTION:
Background

Hyperekplexia, also known as hereditary startle disease or stiff baby syndrome, is a rare neurogenetic non-epileptic disorder characterized by exaggerated persistent startle response and neonatal hypertonia to unexpected auditory, somatosensory and visual stimuli. Startle responses and generalized muscle stiffness both gradually subside during the first months of life. Pathological startle responses can remain throughout adulthood resulting in unprotected falls and injury.

Hereditary hyperekplexia has been identified in 70 pedigrees, most of them being characterized by the major form. Some occasional occurrence of the minor form was described in rare families, but its presence may remain clinically undetected.

The clinical diagnosis of the major form of hyperekplexia needs three mandatory features:

1. Generalized stiffness after birth normalizing during the first years of life
2. Excessive startling to an unexpected stimulus, particularly auditory, present from birth and remaining throughout life
3. Generalized stiffness after a startle reflex that lasts a few seconds Five genes are associated with hyperekplexia, the disease being caused by mutations in the genes encoding different subunits of the inhibitory postsynaptic glycine receptor GLRA1 and GLRB. Additionally defects in the presynaptic glycine transporter gene (SLC6A5) have been recently identified in human hyperekplexia. GPHN, encoding the glycinergic clustering molecule gephyrin, and ARHGEF9, an X-linked gene encoding collybistin, are each associated with one known case of hyperekplexia.

The glycine receptor is a member of the pentameric ligand-gated ion channel family. The receptor is a membrane-embedded protein that contains an integral Cl- -selective pore. The glycine receptor is the major determinant of inhibitory neurotransmission in the retina, spinal cord and brainstem.

Inhibitory synaptic transmission in the spinal cord dorsal horn use GABA and glycine as their principle fast neurotransmitters. Both of them open the Cl- -channels, which induce postsynaptic hyperpolarisation and impairs the propagation of excitatory potentials on dendrites of neurons. Immunofluorescence studies have revealed abundant glycinergic innervations in the dorsal horn, site attributed to the long standing gate control theory of pain. According to this model, inhibitory GABAergic and glycinergic interneurons in the superficial spinal dorsal horn are key components in the control of pain transmission from the periphery to the brain. The model states that a non-painful stimulation is felt as non painful as long as the synaptic GABAergic and glycinergic inhibition remains intact.

Pharmacological blockade of GABAergic and/or glycinergic neurotransmission in the dorsal horn mimics many symptoms of inflammatory and neuropathic pain. Additionally, a loss of synaptic inhibition in the dorsal horn occurs in animal models of experimental pain. This is difficult to prove experimentally in humans, although studies on nociceptive long term potentiation suggest that loss of inhibitory interneurons in the dorsal horn may have a role in the development of chronic pain in patients.

Objective

The aim of this study is to evaluate for the first time in humans whether symptomatic mutations in the glycinergic system affect central pain processing. Positive results would be suggestive for an important role of the glycinergic system in pain modulation and would therefore stimulate further developments for the pharmacological modulation of human pain syndromes.

Methods

Design Assessment of pain thresholds in consecutive hyperekplexia patients and a group of sex and age-matched healthy volunteers.

Subjects We will test consecutive patients with one of the five mutations cited in the introduction. Patients will receive a compensation of 150 Swiss Francs for their participation, plus reimbursement of travel costs.

23 hyperekplexia patients will be recruited. Once the testing of these patients is completed, 45 healthy age and sex-matched controls will be enrolled.

Treatment with a GABA-agonist (mainly clonazepam) will not be discontinued for safety reasons .

Pain tests:

Pressure pain detection threshold (primary outcome) Electric pain detection threshold to single cutaneous and temporal summation to repeated electrical stimulation Heat and cold pain detection, conditioned pain modulation

ELIGIBILITY:
Inclusion Criteria:

* Hyperekplexia
* GLRA1
* GLRB
* SCLA5
* GPHN
* Gephyrin
* ARHGEF9

Exclusion Criteria

* Age below 7 years
* Pregnancy
* Breast feeding
* Ongoing medication
* Cognitive impairment

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pressure pain detection threshold measured in kPA, measured with electronic pressure algometer applied at the centre of the pulp of the 2nd toe | Within 0 to 33 seconds after the beginning of the stimulation
  Pain detection thresholds will be measured with an electronic pressure algometer applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed.

SECONDARY OUTCOMES:
Electric pain reflex, as measured with electromyography from the biceps femoris and the rectus femoris muscles | Within 50 to 150 ms after the beginning of stimulation
  Electromyographic (EMG) reflex responses to electrical stimulation will be recorded from the middle of the biceps femoris and the rectus femoris muscles (Ag/AgCl-electrodes). A 25 ms, train-of-five, 1 ms, square-wave impulse (perceived as a single stimulus), will be delivered. The current intensity will be increased from 1 mA in steps of 1 mA until: 1) a biceps femoris reflex with an amplitude exceeding 20 mV for at least 10 ms in the 50-150 ms post-stimulation interval will be detected (single stimulus reflex threshold); and 2) a pain sensation will be evoked (single stimulus pain threshold).
Heat and cold pain detection thresholds, as measured with a thermode in degrees Celsius | Within 0 to 14 seconds after the beginning of the stimulation
  A thermode will be applied to the skin. The temperature of the thermode will be continuously increased from 30 ºC to a maximum of 50.5 ºC at a rate of 1.5 ºC/s. Pain detection threshold is defined as for pressure stimulation. The subjects are instructed to press a button when this point is reached. For cold stimulation, the temperature of the thermode will be continuously decreased from 30 ºC to a minimum of 0 ºC at a rate of 1.5 ºC/sec. Pain detection threshold is defined as for pressure stimulation. The subjects are instructed to press a button when this point is reached.
Ice water pain threshold of the hand as measured in seconds the hand was left in the water, measured with ice water container | Within 0 to 2 minutes after the beginning of the stimulation
  The device consists of a container separated into an outer and an inner part by a mesh screen. The mesh screen prevents direct contact between the ice (placed in the outer part) and the hand of the subject (placed in the inner part). The water is regularly mixed to maintain the temperature in the inner part near to 0°C. The subject places his hand, wide open and to the wrist, into the inner part of the container. He is asked to keep it in the water until he feels an intolerable sensation of pain and is forced to remove his hand from the container, in any case for a maximum time of 2 min.
Pressure pain detection threshold measured in kPA, measured with electronic pressure algometer applied at the centre of the pulp of the 2nd toe | At the end of the experiment, expected to be after 30 minutes on average
  Pain detection thresholds will be measured with an electronic pressure algometer applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, Prof., Study Chair — Dep. of Anesthesia and Pain medicine, Bern University Hospital
Locations (1):
- Dep. of Anesthesia and Pain medicine, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Zhou L, Chillag KL, Nigro MA. Hyperekplexia: a treatable neurogenetic disease. Brain Dev. 2002 Oct;24(7):669-74. doi: 10.1016/s0387-7604(02)00095-5. PMID 12427512
- [Background] Andermann F, Keene DL, Andermann E, Quesney LF. Startle disease or hyperekplexia: further delineation of the syndrome. Brain. 1980 Dec;103(4):985-97. doi: 10.1093/brain/103.4.985. PMID 6777025
- [Background] Praveen V, Patole SK, Whitehall JS. Hyperekplexia in neonates. Postgrad Med J. 2001 Sep;77(911):570-2. doi: 10.1136/pmj.77.911.570. PMID 11524514
- [Background] Muller F, Heinke B, Sandkuhler J. Reduction of glycine receptor-mediated miniature inhibitory postsynaptic currents in rat spinal lamina I neurons after peripheral inflammation. Neuroscience. 2003;122(3):799-805. doi: 10.1016/j.neuroscience.2003.07.009. PMID 14622922